CLINICAL TRIAL: NCT01275690
Title: Noninvasive Cardiac Output Measurements in Patients With Pulmonary Hypertension Undergoing Right Heart Catheterization With Acute Vasodilator Testing
Status: Withdrawn | Type: Observational
Why Stopped: The PI closed this study and went to another institution.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 10-179-B
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Hypertension
Keywords: cardiac; pulmonary hypertension; To determine the accuracy of a noninvasive method of measuring cardiac output as compared to the standard invasive approach in patients with PH
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- subjects with PH undergoing right heart catheterization

SUMMARY:
Subjects in this study have been diagnosed with pulmonary hypertension (PH) and their doctors have referred them for a right heart catheterization (RHC). Heart catheterization involves inserting an IV (a needle with a small tube) into a vein in the neck. A long, narrow tube, called a catheter, is guided through the IV into the blood vessel and guided to the heart (sometimes this procedure can be done through a vein in the groin instead). Once the catheter is in place, small instruments can be inserted into the catheter to measure the pressures in different areas of the heart. These measurements can help the doctor diagnose possible problems with the heart functioning.

The purpose of this study is to evaluate the measurements provided by a device, called Noninvasive Cardiac Output Monitoring (NICOM). The NICOM device is non-invasive which means the investigators do not have to go inside the body to obtain the heart pressure measurements. While the device has been approved for use in any patient, it remains possible that patients with PH will have differences in the way the device calculates measurements. In this study, the investigators will compare the in-the-body (right heart catheterization) measurements to the non-invasive, outside-body measurements provided by the NICOM device to evaluate any differences.

The NICOM device is approved by the US Food and Drug Administration (FDA) to measure heart pressures. This device is usually used when a patient can't undergo a right heart catheterization. In this study, the investigators are using the device to gather heart pressure measurements for research during the right heart catheterization procedure that is scheduled as part of the patients' normal, routine care. The research data is being used to devise better, less invasive ways to assess disease severity, track disease progression and evaluate response to therapy. The NICOM device is made by Cheetah Medical.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and up
* have Pulmonary Hypertension (PH)
* Scheduled for cardiac catheterization with right heart catheterization and acute vasodilator testing as part of their evaluation of PH

Exclusion Criteria:

* unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll 100 consecutive patients referred to the Pulmonary Hypertension Center and scheduled for cardiac catheterization with right heart catheterization and acute vasodilator testing as part of their evaluation of PH.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
To determine the accuracy of a noninvasive method of measuring cardiac output as compared to the standard invasive approach using thermodilution in patients with pulmonary hypertension | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Archer, MD, Principal Investigator — University of Chicago